CLINICAL TRIAL: NCT06576401
Title: A Phase1 Study to Characterize Mass Balance Of [14C] HDM1002 in Chinese Healthy Subjects
Brief Title: A Study To Characterize Mass Balance Of [14C] HDM1002 in Chinese Healthy Subjects
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou Zhongmei Huadong Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HDM1002-104
Record Dates: First submitted 2024-08-20; First posted 2024-08-28 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2024-09

CONDITIONS: Healthy Adult Subject
Keywords: HDM1002; Glucagon-Like Peptide-1 Receptor Agonists

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C] HDM1002 (Experimental): A single dose of HDM1002 and [14C] HDM1002 administered orally.
  Interventions: Drug: [14C] HDM1002

INTERVENTIONS:
Drug: [14C] HDM1002 — Administered orally

SUMMARY:
In this study, a single dose of [14C] radiolabelled HDM1002 will be administered orally. The main purpose of this study is to find out how much of HDM1002 and its metabolites pass from blood into urine and feces, and characterize the metabolic profile and routes of excretion of oral [14C] HDM002.

ELIGIBILITY:
Inclusion Criteria:

1. Male, healthy adult;
2. Age of 18 to 45 years old (both inclusive);
3. Body mass index (BMI) between 19.0- 32.0 kg/m2 (both inclusive) and body weight no less than 50.0 kg.

Exclusion Criteria:

1. Clinically significant diseases at the time of screening;
2. History or family history of medullary thyroid carcinoma, thyroid C-cell hyperplasia, or multiple endocrine neoplasia type 2 (MEN2), or calcitonin ≥ 35 ng/L during the screening period;
3. History of chronic pancreatitis or acute pancreatitis within 3 months prior to screening;
4. History of acute cholecystitis attack within 3 months prior to screening;
5. Participant judged by investigator has dysphagia, diseases or conditions that affect gastric emptying or affect the absorption of nutrients in the gastrointestinal tract, such as bariatric surgery or other gastrectomy, irritable bowel syndrome, dyspepsia, etc.;
6. Any of the following: habitual constipation or diarrhea, hemorrhoids or accompanied by perianal disease, irritable bowel syndrome, inflammatory bowel disease, etc;
7. Use of any prescription medication, over-the-counter medication, Chinese herbal medicine or food supplement within 14 days or 5 half-lives (whichever is longer) prior to the screening period;
8. Patients with any abnormal and clinically significant examinations in given comprehensive physical examination;
9. History of drug abuse (e.g., morphine, ketamine, tetrahydrocannabinolic acid, metham phetamine, methylenedioxyamphetamine, cocaine) or positive urine drug test during the screening period;
10. Positive for hepatitis B surface antigen or E antigen, hepatitis C virus antibody IgG (Anti-HCV IgG), human immunodeficiency virus antigen/antibody combination test (HIV-Ag/Ab) and Treponema pallidum antibody during the screening period.
11. Engaged in working conditions requiring long-term exposure to radioactivity; or significant radioactive exposure ( ≥ 2 CT chest/abdomen tests, or ≥ 3 all other types of X-rays test) within 1 year prior to the trail, or participated in radio-label trails;

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-08-27 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Total recovery of HDM1002 radioactivity in urine and feces, following oral administration of [14C] HDM1002 | Predose up to Day 11 after administration of [14C] HDM1002
  Total recovery of radioactivity in urine and feces, and both routes combined expressed as a percentage of the total radioactive dose administered
Metabolite profiling/identification in plasma, urine, and feces | Predose up to Day 11 after administration of [14C] HDM1002
  Metabolic profiling/identification and determination of relative abundance of [14C]PF-06882961 and the metabolites of [14C] HDM1002 in plasma, urine, and feces.
Plasma and whole blood AUC[0-t] of radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Area under the curve from time 0 to t hour
Plasma and whole blood AUC[0-∞] of radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Area under the curve from time 0 hour to ∞
Plasma and whole blood Cmax of radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Maximum observed concentration
Plasma and whole blood Tmax of radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Time to maximum plasma concentration
Plasma and whole blood t1/2 of radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter: Half life
Plasma and whole blood CL/F of radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Apparent Clearance
Plasma and whole blood Vz/F of radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Apparent volume of distribution
Percentage of plasma HDM1002 and metabolites in total plasma radioactivity | Predose up to Day 11 after administration of [14C] HDM1002
  Percentage of plasma HDM1002 AUC in total plasma radioactivity AUC

SECONDARY OUTCOMES:
Plasma AUC[0-t] of HDM1002 and metabolites | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Area under the curve from time 0 to t hour
Plasma AUC[0-∞] of HDM1002 and metabolites | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Area under the curve from time 0 hour to ∞
Plasma Cmax of HDM1002 and metabolites | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Maximum observed concentration
Plasma Tmax of HDM1002 and metabolites | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Time to maximum plasma concentration
Plasma t1/2 of HDM1002 and metabolites | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter: Half life
Plasma CL/F of HDM1002 and metabolites | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Apparent Clearance
Plasma Vz/F of HDM1002 and metabolites | Predose up to Day 11 after administration of [14C] HDM1002
  PK parameter : Apparent volume of distribution
Adverse events (AEs) | Predose up to Day 11 after administration of [14C] HDM1002
  Number of subjects reporting AEs

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China